CLINICAL TRIAL: NCT04179188
Title: Impact of Bariatric Surgery in Obese Patients With and Without Obstructive Sleep Apnea Syndrome - COLOSS
Brief Title: Impact of Bariatric Surgery in Obese Patients With and Without Obstructive Sleep Apnea Syndrome
Acronym: COLOSS
Status: Recruiting | Type: Observational
Sponsor: Ramsay Générale de Santé (Other)
Collaborators: Dr CODRON (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2019-A00832-55
Record Dates: First submitted 2019-11-25; First posted 2019-11-27 (Actual); Last update posted 2019-11-27 (Actual); Status verified 2019-11

CONDITIONS: Obesity; Bariatric Surgery Candidate; Apnea, Obstructive
Keywords: obesity; Bariatric Surgery; Obstructive Sleep Apnea
MeSH Terms: conditions — Obesity; Sleep Apnea, Obstructive | interventions — Bariatric Surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Bariatric OSA Group: Bariatric surgery plannified intervention patient with obstructive sleep Apnéa
  Interventions: Procedure: Bariatric surgery
- Bariatric without OSA Group: Bariatric surgery plannified intervention patient without obstructive sleep Apnéa
  Interventions: Procedure: Bariatric surgery

INTERVENTIONS:
Procedure: Bariatric surgery — Classical Bariatric surgery (ring, Sleeve gastrectomy or Bypass)

SUMMARY:
It has been shown to date that obesity is associated with increased mortality and that weight loss significantly improves cardiovascular risk factors. Among patients receiving bariatric surgery, 30-90% have moderate to severe obstructive sleep apnea (OSA) syndrome. Given the strong associations between OSA and cardiometabolic comorbidities, this project is based on the hypothesis of a lower improvement of cardiovascular risk factors and a higher number of post-surgical complications in OSAS patients.

DETAILED DESCRIPTION:
It has been shown to date that obesity is associated with increased mortality and that weight loss significantly improves cardiovascular risk factors.

Bariatric surgery is now the most effective intervention for the long-term treatment of obesity and its complications. Among patients receiving bariatric surgery, 30-90% have moderate to severe obstructive sleep apnea (OSA) syndrome. The progressive loss of weight contributes to the regression of the symptoms related to OSA. Observational studies have shown that bariatric surgery can rapidly improve glycemic control and cardiovascular risk factors with a significantly higher remission rate of hypertension and dyslipidemias than in the non-surgical group. Given the strong associations between OSA and cardiometabolic comorbidities, this project is based on the hypothesis of a lower improvement of cardiovascular risk factors and a higher number of post-surgical complications in OSAS patients.

ELIGIBILITY:
Inclusion Criteria:

* Patient, male or female, aged over 18
* Patient in preparation for bariatric surgery (ring, Sleeve gastrectomy or Bypass) in the center CELIOBE.
* Patient affiliated with social security or beneficiary of such a scheme
* Patient having signed the free and informed consent

Exclusion Criteria:

* Patient who has already had bariatric surgery (ring, sleeve gastrectomy or bypass).
* Patient already receiving CPAP treatment for sleep apnea syndrome.
* Patients with pathology indicating the use of CPAP in self-guided mode (heart failure with altered ejection fraction) for patients diagnosed with OSAS
* Patient likely, in the opinion of the investigator, not to be cooperative or respectful of the obligations inherent to participation in the study
* Patient suffering from mental pathology does not make possible the collection of a consent.
* Protected patient: major under guardianship, curatorship or other legal protection, deprived of liberty by judicial or administrative decision
* Pregnant, lactating or parturient woman
* Patient hospitalized without consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient in preparation for bariatric surgery in the center CELIOBE
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2019-10-09 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Hypertension | 1 year
  The primary endpoint is the measurement of Systolic and Diastolic Blood Pressure.

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital privé La Louvière, Lille, Haut de France, France

IPD SHARING:
Plan to Share IPD: Undecided